CLINICAL TRIAL: NCT07118644
Title: Microbiote's Evolution After Use of Nitrous Oxide on Pediatric Patient Needing Airway Samples
Acronym: MicroNO
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 29BRC23.0238; 2024-518197-14-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-04; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Respiratory Ilness; Children
Keywords: Lung microbiota; MEOPA; Infant
MeSH Terms: interventions — Meopa

STUDY DESIGN:
Intervention Model Description: This is an exploratory, controlled, open-label, prospective, monocentric clinicobiological case control study. Each case is its own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case (Experimental): Induced sputum with MEOPA
  Interventions: Drug: MEOPA
- Control (Other): Standard induced sputum
  Interventions: Other: Standard induced sputum

INTERVENTIONS:
Drug: MEOPA — Induced sputum with be performed by trained physiotherapist using hypertonic saline aerosol and salbutamol. MEOPA will be used for nebulization. MEOPA is a gas with analgesic, amnesic and anxiolytic properties.
  Arms: Case
Other: Standard induced sputum — Induced sputum with be performed by trained physiotherapist using hypertonic saline aerosol and salbutamol. Oxygen will be used for nebulization.
  Arms: Control

SUMMARY:
The objective of this study is to determine whether the use of MEOPA alters the composition of respiratory microbiota collected by induced sputum in children requiring respiratory sampling for suspected lower respiratory tract infection.

Children aged 3 months to 8 years and they requiring ECBC sampling in routine practice.

DETAILED DESCRIPTION:
This is an exploratory, controlled, open-label, prospective, monocentric clinicobiological case control study. Each case is its own control. A sample will be taken without MEOPA and then with MEOPA.

The Infants will be included after written informed consent will be obtained from the patients' parents or legally authorized representatives. Cytological and microbiological analyses are carried out on each sample.

ELIGIBILITY:
Inclusion Criteria:

* Children aged from 3 months to 8 years old
* Patients requiring ECBC in routine practice: acute respiratory distress with suspected bacterial respiratory infection (superinfected bronchiolitis or asthma attack, suspected pneumonia) and severe asthma assessment
* Child unable to expectorate effectively
* Free, informed and written consent of the minor patient's legal guardians;
* Enrolled in the social security system.

Exclusion Criteria:

1. Contraindication of MEOPA :

   * Patients requiring 100% oxygen ventilation
   * Intracranial hypertension
   * Altered state of consciousness preventing cooperation
   * Any condition where air is trapped inside the body and expansion could be dangerous (cranial and/or maxillofacial trauma, pneumothorax, emphysema, gas embolism, following recent scuba diving, decompression sickness following gas encephalography, during middle ear/internal ear or sinus surgery, abdominal gas distension, when air is injected into the epidural space during epidural anesthesia, if the patient has received ophthalmic gas (SF6, C3F8, C2F6) used in eye surgery for as long as the gas bubble persists and up to 3 months afterwards)
   * Known, unsubstituted vitamin B12 or folic acid deficiency
   * Recent, unexplained neurological abnormalities
2. Contraindications to induced expectoration :

   * Clinical instability not conducive to induced expectoration (at practitioner's discretion)
   * Severe respiratory insufficiency,
   * Severe spasticity.
   * Hemoptysis
   * Decompensated heart failure
   * Contraindication of hypertonic saline :
   * Hypersensitivity of the bronchial system to hypertonic sodium chloride solutions.
   * Hemoptysis
   * Contraindication to the use of Salbutamol :
   * Hypersensitivity to any of the constituents of salbutamol-based pressurized or inhaled products.
   * Intolerance to salbutamol-based pressurized or inhaled products (coughing or bronchospasm occurring immediately after inhalation of the product).
   * Contraindication of the maneuver performed by the physiotherapist: bullous emphysema, confirmed hiatal or diaphragmatic hernia and rib fragility.
3. Patient with minor parent(s)
4. Uncooperative child
5. Antibiotic therapy administered within the previous 24 hours.

Ages: 3 Months to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-06 (Estimated); Study Completion 2027-09-06 (Estimated)

PRIMARY OUTCOMES:
α and β diversities | Day 1
  These outcomes will be calculated from ASV table obtained from 16S metagenomic analysis.

SECONDARY OUTCOMES:
Children anxiety | Day 1
  mYPAS-SF (Modified Yale Preoperative Anxiety Scale, short version) total score before and after each induced sputum. Score between 4 and 18 (18 is the maximum level of anxiety)
Feeling of physiotherapist about the child's behaviour | Day 1
  Likert scale after each induced sputum
Feeling of parent(s) about the child's behaviour | Day 1
  Visual Analogue Scale (VAS) after each induced sputum
Sputum induced adverse events | Day 5
  Number of adverse events related to induced expectoration
Specimen quality | Day 1
  Murray and Washington cytological score (good quality specimen: score ≥ 3; poor quality specimen: score < 3)
Search for microbiota mismatch with or without meopa | Day 1
  The criterion is defined by an expert opinion indicating whether the results of the examinations are concordant, or discordant against MEOPA or discordant in favor of MEOPA
Bacterial taxa | Day 1
  Bacterial taxa is identified by 16S v3-v4 targeted metagenomics.
Adverse Events | Day 5
  Number of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Brest, University Hospital, Brest, France